CLINICAL TRIAL: NCT00459563
Title: A Randomized Placebo-controlled Double Blinded Trial to Evaluate Cholecalciferol (Vitamin D3) and Calcitriol Treatment on Reducing Blood Pressure in Middle Aged Adults With Stage I Hypertension and Vitamin D Deficiency
Brief Title: Vitamin D and Blood Pressure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Vin Tangpricha, Staff Physician, Atlanta VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 648-2006; VAMC Atlanta R&D AREF 283001
Record Dates: First submitted 2007-04-10; First posted 2007-04-12 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
Keywords: vitamin D; blood pressure; hypertension; Vitamin D insufficient; Systolic blood pressure between 130 and 150 mmHg
MeSH Terms: conditions — Hypertension | interventions — Vitamin D; Calcitriol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cholecalciferol (Active Comparator): Cholecalciferol
  Interventions: Drug: Vitamin D
- Calcitriol (Active Comparator): Calcitriol
  Interventions: Drug: calcitriol

INTERVENTIONS:
Drug: Vitamin D — 200,000 IU once weekly for 3 weeks (600,000 IU total dose)
  Arms: Cholecalciferol
Drug: calcitriol — calcitriol 0.5 mcg twice a day for 1 week
  Arms: Calcitriol
Drug: Placebo — Placebo once a week for 3 weeks
  Arms: Placebo

SUMMARY:
Vitamin D is a natural nutrient in normal daily diet. It can also be made in the skin after exposure to sunlight and is essential for maintaining normal calcium balance. One past study has suggested that vitamin D may be helpful for blood pressure. This study will test whether pills containing cholecalciferol (a form of vitamin D) or calcitriol (the active form of vitamin D) can treat high blood pressure. The investigators plan to enroll up to 80 subjects at the Atlanta VA Medical Center. Participation in the study is expected to last up to 4 weeks. Subjects will be assigned to cholecalciferol, calcitriol or placebo). A 24-hour blood pressure monitor will be worn at the beginning and end of the study to determine blood pressure changes. Renin, PTH, angiotensin-II, and aldosterone levels will also be measured at the beginning and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over the age of 18
* Vitamin D levels between 10 and 30 ng/ml
* Systolic blood pressure between 130 and 150 mmHg

Exclusion Criteria:

* Current use of anti-hypertensive medication
* Inability to understand the consent form
* Inability to return ABP monitor within 24-48 hours after visit
* Alcohol dependence
* Diagnosis of chronic kidney disease
* History of heart disease
* History of stroke
* Inability to comply with study protocol
* Current treatment for cancer
* Narcotic dependence
* Current use of greater than 2000 IU of vitamin D
* Pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 3 Weeks
25(OH)D | 3 weeks

SECONDARY OUTCOMES:
Parathyroid hormone | 3 weeks
Renin | 3 weeks
Aldosterone | 3 weeks
Angiotensin II | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vin Tangpricha, MD/PhD, Principal Investigator — Emory University/VAMC; Suzanne E Judd, MPH, Study Director — Emory University
Locations (1):
- VAMC, Decatur, Georgia, United States